CLINICAL TRIAL: NCT06661798
Title: Evaluation of Changes in Mental Foramen Blood Flow After Orthognathic Surgery Using Ultrasound
Brief Title: Evaluation of the Mental Foramen After Surgery Via Ultrasonography
Acronym: Blood flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Elifhan Alagoz, Assistant Professor, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 27.02.2024-E.142577
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-10

CONDITIONS: Orthognathic Surgery
Keywords: Mental foramen; orthognathic surgery; blood flow; ultrasonography
MeSH Terms: interventions — Orthognathic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orthognathic surgery (Other): Patients who have reached skeletal maturity, have skeletal Class II or Class III malocclusion, and are indicated for orthognathic surgery due to malocclusion complaints
  Interventions: Procedure: orthognathic surgery; Procedure: USG examination; Procedure: Subjective evaluation - Neuro-sensitivity tests

INTERVENTIONS:
Procedure: orthognathic surgery — Mandibular setback, Maxillary advancement, Bilateral sagital split osteotomy
Procedure: USG examination — Comparison of blood flow in the mental foramen before and 1week, 1 month and 3 month after orthognathic surgery using ultrasound examination
Procedure: Subjective evaluation - Neuro-sensitivity tests — Direction determination, two-point separation, pinprick, and brush tests, along with neurosensitivity VAS and pressure VAS, were applied to the patients. These tests were performed before surgery (T0), seven days after surgery (T1), one month after surgery (T2), and three months after surgery (T3).

SUMMARY:
Objective: This study aims to detect changes in blood flow in the mental foramen after surgery compared to before orthognathic surgery.

Materials and Methods: This study will include a total of 16 patients, aged between 18-60, who were planned for orthognathic surgery due to malocclusion complaints. Patients will be evaluated clinically and radiologically before surgery, 1 week, 1 month, and 3 months after the surgery. Panoramic radiographs will be taken before surgery and 3 months after surgery, and a fractal analysis of the ROI area determined distal to the mental foramen will be performed. Pain will be scored from 1 to 5 using the Pinprick test before surgery, 1 week, 1 month, and 3 months after surgery, while pressure and neurosensitivity will be scored using VAS. Neurosensory evaluation will be performed using two-point discrimination (dividing the area between the lower lip and chin into 9 regions), and left-right discrimination will be checked using the brush test. Blood flow in the mental foramen will be evaluated using ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old,
2. Patients who have reached skeletal maturity,
3. Patients under 60 years old,
4. Patients with skeletal Class II malocclusion indicated for orthognathic surgery,
5. Patients with skeletal Class III malocclusion indicated for orthognathic surgery,
6. Those who are willing to participate in the study

Exclusion Criteria:

1. Patients with a systemic disease,
2. Patients under 18 years old,
3. Patients who have not completed their growth and development,
4. Patients over 59 years old,
5. Patients using neurological and psychiatric medications,
6. Patients who have previously undergone surgery or experienced trauma in the mandibular region,
7. Patients with neurosensory dysfunction in the inferior alveolar nerve before surgery,
8. Pregnant individuals or those suspected of being pregnant,
9. Any local or systemic condition that may contraindicate general anesthesia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Changes in blood flow in the mental foramen after orthognathic surgery | From enrollment to 3 months after the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No